CLINICAL TRIAL: NCT00684125
Title: Evaluation of Different Strategies of Pericardial Drainage After Aortic Valvular Surgery: A Prospective Randomized Trial
Brief Title: Evaluation of Different Strategies of Pericardial Drainage After Aortic Valvular Surgery
Acronym: Blake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Philippe Demers M.D., M.Sc., FRCSC, Montreal Heart Institute - Cardiac surgeon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICM 07-934
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Pericardial Effusion; Late Cardiac Tamponade; Surgical Reintervention
Keywords: late cardiac tamponade
MeSH Terms: conditions — Pericardial Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): mediastinal drainage will be accomplished using a 28F or 32F chest tube in the anterior mediastinum and a 19F Blake drain located in the posterior pericardial cavity.
  Interventions: Device: Blake Drains (Blake drain, Ethicon USA)
- 2 (Active Comparator): mediastinal drainage will be accomplished using two 28F or 32F chest tubes located in the anterior mediastinum.
  Interventions: Device: Standard mediastinal drainage

INTERVENTIONS:
Device: Blake Drains (Blake drain, Ethicon USA) — 19F Blake drain located in the posterior pericardial cavity
  Other Names: Blake drain: prolonged mediastinal drainage
  Arms: 1
Device: Standard mediastinal drainage — Mediastinal drainage will be accomplished using 28F or 32F chest tube located in the anterior mediastinum
  Other Names: mediastinal drainage
  Arms: 2

SUMMARY:
The incidence of pericardial effusion and late cardiac tamponade after aortic and valvular surgery is higher than after other cardiac surgical procedures. The aim of this study is to evaluate the clinical safety and efficacy of prolonged mediastinal drainage using small, soft silastic drains (Blake drain, Ethicon USA) versus conventional mediastinal drainage using large chest tubes. A prospective randomized trial.

DETAILED DESCRIPTION:
The incidence of pericardial effusion and late cardiac tamponade after aortic and valvular surgery is higher than after other cardiac surgical procedures. The aim of this study is to evaluate the clinical safety and efficacy of prolonged mediastinal drainage using small, soft silastic drains (Blake drain, Ethicon USA) versus conventional mediastinal drainage using large chest tubes. Patients undergoing aortic and / or valvular surgery will be randomized in two groups. In group A, mediastinal drainage will be accomplished using a 28F or 32F chest tube in the anterior mediastinum and a 19F Blake drain located in the posterior pericardial cavity. In group B, mediastinal drainage will be accomplished using two 28F or 32F chest tubes located in the anterior mediastinum. In both groups, conventional chest tubes will be removed on the first postoperative day, while patients in the group A will have prolonged drainage using the Blake drain until output is less than 50 ml over 24 hour. Patients will be followed during their postoperative course for occurrence of significant pericardial effusion as detected on routine echocardiogram and late cardiac tamponade requiring reintervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 90 years old, undergoing either surgery of the ascending and/or transverse aorta, or surgery of the mitral and/or aortic valves
* Availability for follow-up at the Montreal Heart Institute Exclusion criteria

Exclusion Criteria:

* Emergency surgery
* Unavailability for follow-up at the Montreal Heart Institute

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Any pericardial effusion of 15 mm or more as measured on postoperative transthoracic echocardiogram on day 5 and late cardiac tamponade requiring surgical reintervention. | Day 5 - post surgery

SECONDARY OUTCOMES:
Total volume of mediastinal drainage. Pain intensity on postoperative days 1 to 5. Incidence of postoperative atrial fibrillation Drain-associated infection or any other drain-associated adverse event. | Days 1 or till discharge - post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe Demers, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Eryilmaz S, Emiroglu O, Eyileten Z, Akar R, Yazicioglu L, Tasoz R, Kaya B, Uysalel A, Ucanok K, Corapcioglu T, Ozyurda U. Effect of posterior pericardial drainage on the incidence of pericardial effusion after ascending aortic surgery. J Thorac Cardiovasc Surg. 2006 Jul;132(1):27-31. doi: 10.1016/j.jtcvs.2006.01.049. PMID 16798298
- [Background] Agati S, Mignosa C, Gitto P, Trimarchi ES, Ciccarello G, Salvo D, Trimarchi G. A method for chest drainage after pediatric cardiac surgery: a prospective randomized trial. J Thorac Cardiovasc Surg. 2006 Jun;131(6):1306-9. doi: 10.1016/j.jtcvs.2006.02.013. PMID 16733162
- [Background] Ege T, Tatli E, Canbaz S, Cikirikcioglu M, Sunar H, Ozalp B, Duran E. The importance of intrapericardial drain selection in cardiac surgery. Chest. 2004 Nov;126(5):1559-62. doi: 10.1378/chest.126.5.1559. PMID 15539727
- [Background] Obney JA, Barnes MJ, Lisagor PG, Cohen DJ. A method for mediastinal drainage after cardiac procedures using small silastic drains. Ann Thorac Surg. 2000 Sep;70(3):1109-10. doi: 10.1016/s0003-4975(00)01800-2. PMID 11016389
- [Background] Kuvin JT, Harati NA, Pandian NG, Bojar RM, Khabbaz KR. Postoperative cardiac tamponade in the modern surgical era. Ann Thorac Surg. 2002 Oct;74(4):1148-53. doi: 10.1016/s0003-4975(02)03837-7. PMID 12400760
- [Background] Shah A, van den Brink A, de Mol B. Raised international normalized ratio: an early warning for a late cardiac tamponade? Ann Thorac Surg. 2006 Sep;82(3):1090-1. doi: 10.1016/j.athoracsur.2006.01.035. PMID 16928545
- [Derived] Moss E, Miller CS, Jensen H, Basmadjian A, Bouchard D, Carrier M, Perrault LP, Cartier R, Pellerin M, Demers P. A randomized trial of early versus delayed mediastinal drain removal after cardiac surgery using silastic and conventional tubes. Interact Cardiovasc Thorac Surg. 2013 Jul;17(1):110-5. doi: 10.1093/icvts/ivt123. PMID 23575759